CLINICAL TRIAL: NCT03977558
Title: The Effect of Canola Oil Consumption on the Selected Cardiometabolic Parameters in a Group of Shift Workers
Brief Title: Health Effect of Canola Oil Consumption in Shift Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Kuleta-Koberska, Principal Investigator, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IoHNaD
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Shift-Work Related Sleep Disturbance; Metabolic Syndrome; Diet Modification; Work-Related Condition
Keywords: Shift Work; Night Work; Rotating Shift Work; Metabolic Syndrome; Diet Therapy; Canola oil; Fatty Acids; Cardiometabolic parameters
MeSH Terms: conditions — Metabolic Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Isocaloric diet, based on individual energy requirements calculated from indirect calorimetry and physical activity adjustment Participants will be asked to eat daily ~50g canola oil
  Interventions: Behavioral: Intervention group
- Control group (Active Comparator): Standard dietary advice that is used as current best practice in the treatment of lipid disturbances of European Society of Cardiology and European Atherosclerosis Society (ESC/EAS) Guidelines for the management of dyslipidemias)
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — Isocaloric diet including ~50g canola oil
  Arms: Intervention group
Behavioral: Control group — ESC/EAS Guidelines for the management of dyslipidemias
  Arms: Control group

SUMMARY:
Shift work is associated with a higher risk of the development of cardiometabolic syndrome (CMtS) than in people working only during the day. One of the factors predisposing to the development of the CMtS in shift workers is an inappropriate composition of their diet. It was observed that the shift workers diet is characterized by a higher intake of saturated fatty acids (SFA) and a lower consumption of unsaturated fatty acids. One potential way to reduce the risk of CMtS in this study group seems to be a modification of their everyday diet by excluding the products of animal origin (e.g. butter) with simultaneously including vegetable oils (i.e. canola oil). The aim of the study is to evaluate the effect of replacement in the everyday diet of saturated fats (butter) with unsaturated fats (canola oil-based spread and canola oil added to main meals) in centrally obese shift workers on changes in body weight and body composition parameters as well as on changes in CMtS markers.

DETAILED DESCRIPTION:
The study was designed as a randomized clinical trial to investigate the effects of the dietary intervention with moderate in fat content (~35% energy as fat) for 12 weeks on the improvement of cardiometabolic risk factors in centrally obese shift workers. Forty centrally obese shift workers (waist circumference ≥94 cm) were randomized (1:1) to the experimental group (n = 20) or the control group (n = 20). Eligibility criteria included: aged between 30-60 years, working rotating shifts for at least 5 years and working night shifts minimum five times a month. Excluded criteria was described in the point "Eligibility". Written informed consent was obtained from all of the participants, and the local ethic committee approved the study. The dietary intervention was mainly based on the simple rearrangement of shift workers' diets by replacing food items including SFA (e.g. butter) with those being sources of unsaturated fatty acids (UFA), mainly canola oil (given to the diet as spread or this oil was added separately to main meals)

ELIGIBILITY:
Inclusion Criteria:

* centrally obese (≥ 94cm) male
* aged between 30-60 years,
* working rotating shifts for at least 5 years and working night shifts minimum five times a month,

Exclusion Criteria:

* diabetes, familial hypercholesterolemia, thyroid and parathyroid diseases, non-specific intestinal diseases, celiac disease, phenylketonuria,
* taking medication for lowering blood lipids such as statins,
* weight loss therapy for 3 months before the intervention,
* allergies and intolerances
* consuming high-proof alcoholic beverages (>2 portions/week)

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Waist circumference (WC) | Baseline, 4, 8 and 12 week
  Changes in WC within groups and between groups
HDL-cholesterol (HDL-C) | Baseline, 12 week
  Changes in HDL-C within groups and between groups
LDL-cholesterol (LDL-C) | Baseline, 12 week
  Changes in LDL-C within groups and between groups
Triglycerides (TG) | Baseline, 12 week
  Changes in TG within groups and between groups
Glucose (GLU) | Baseline, 12 week
  Changes in GLU within groups and between groups
Blood pressure (BP) | Baseline, 12 week
  Changes in BP within groups and between groups
Body weight (BW) | Baseline, 4, 8 and 12 week
  Changes in BW within groups and between groups
Fat mass (FM) | Baseline, 4, 8 and 12 week
  Changes in FM within groups and between groups

SECONDARY OUTCOMES:
Insulin (INS) | Baseline, 12 week
  Changes in INS within groups and between groups
High-sensitivity C-reactive Protein (hs-CRP) | Baseline, 12 week
  Changes in hs-CRP within groups and between groups
Cardiotrophin-1 (CT-1) | Baseline, 12 week
  Changes in CT-1 within groups and between groups
Lipase (LPS) | Baseline, 12 week
  Changes in LPS within groups and between groups
Cholinesterase (CHE) | Baseline, 12 week
  Changes in CHE within groups and between groups respectively
Alanine transaminase (ALT) | Baseline, 12 week
  Changes in ALT within groups and between groups
Aspartate transaminase (AST) | Baseline, 12 week
  Changes in AST within groups and between groups
Gamma-glutamyltransferase (GGTP) | Baseline, 12 week
  Changes in GGTP within groups and between groups
Melatonin (MEL) | Baseline, 12 week
  Changes in MEL within groups and between groups
Fatty acids (FA) erythrocyte membranes concentration | Baseline, 12 week
  Changes in FA within groups and between groups
Dietary intake | Baseline, 4, 8, 12 week
  Changes in dietary intake within groups and between groups

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Kuleta-Koberska, Msc, Principal Investigator — Poznan University of Life Sciences
Locations (1):
- Poznan University of Life Science, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No